CLINICAL TRIAL: NCT02434445
Title: Use of Novel Plasma and Urinary Biomarkers to Predict the Development of Hepatorenal Syndrome in Cirrhotic Patients
Status: Recruiting | Type: Observational
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Society of Nephrology (Other)
Responsible Party: Principal Investigator, Dr. Desmond Yat-Hin Yap, Clinical Assistant Professor, The University of Hong Kong
Other Study IDs: UW12342
Record Dates: First submitted 2015-04-30; First posted 2015-05-05 (Estimated); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Hepatorenal Syndrome
MeSH Terms: conditions — Hepatorenal Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — patient's serum and urine samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Hepatorenal syndrome group: Patients with advanced cirrhosis who develope hepatorenal syndrome
- Non-hepatorenal syndrome group: Patients with advanced cirrhosis who do not hepatorenal syndrome

SUMMARY:
This study investigated the use of novel plasma and urinary biomarkers to predicte the development of hepatorenal syndrome in patients with advanced cirrhosis. The biomarkers investigated include plasma cystatin C, plasma NGAL, plasma NAG, plasma IL-18, plasma ADMA, plasma BTP, urinary KIM-1 and urinary LFABP. These biomarkers will be checked in advanced cirrhotic patients who have or have not developed hepatorenal syndrome and compared between the two groups. These biomarkers will also be correlated with the occurence of hepatorenal syndrome.

DETAILED DESCRIPTION:
This study investigated the use of novel plasma and urinary biomarkers to predicte the development of hepatorenal syndrome in patients with advanced cirrhosis. The biomarkers tested include plasma cystatin C, plasma NGAL, plasma NAG, plasma IL-18, plasma ADMA, plasma BTP, urinary KIM-1 and urinary LFABP. These biomarkers will be checked in advanced cirrhotic patients who have or have not developed hepatorenal syndrome and compared between the two groups. These biomarkers will also be correlated with the occurence of hepatorenal syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced cirrhosis (Child's B or C) referred for liver transplantation
* Willing to give informed consent

Exclusion Criteria:

* Patients with co-existing renal diseases

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced cirrhosis (Child's B or C) referred for liver transplantation
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-06-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Hepatorenal syndrome | 12 weeks

SECONDARY OUTCOMES:
Mortality | 6 months
Chronic renal impairment | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Desmond Yap, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong, Hong Kong